CLINICAL TRIAL: NCT06615648
Title: The Effectiveness of the Protection Motivation Theory in Reducing Alcohol-Related Intentions and Behaviours Among Young Adults
Brief Title: Effectiveness of a PMT Intervention to Reduce Alcohol in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Principle Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PMT and Alcohol
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Behavior, Drinking; Alcohol Drinking; Colorectal Cancer Control and Prevention; Healthy Volunteers
Keywords: Protection Motivation Theory; Alcohol; Alcohol Intention; Alcohol Behaviour; Colorectal Cancer; Behaviour Change
MeSH Terms: conditions — Drinking Behavior; Alcohol Drinking; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PMT Information (Experimental): The participant will watch the PMT-video and then complete the associated questionnaires.
  Interventions: Behavioral: PMT
- Non-contact Control (Active Comparator): The participant will watch a non-specific video about coffee and then complete the associated questionnaires.
  Interventions: Behavioral: Non-contact Control

INTERVENTIONS:
Behavioral: PMT — 7-minute PMT intervention video
  Arms: PMT Information
Behavioral: Non-contact Control — 6-minute alternative video
  Arms: Non-contact Control

SUMMARY:
This study will examine the effectiveness of a 7-minute informational video using the threat and coping components of the Protection Motivation Theory (PMT) reduces alcohol intention and behaviour among young Canadian adults. Our aim is to determine whether perceived vulnerability, perceived severity, response efficacy and self-efficacy are associated with goal intentions to reduce drinking alcohol, and whether goals intentions to reduce alcohol drinking are associated with actual reductions in alcohol use among this population. Participants will be randomized to view either a specific PMT-video or a non-specific video on coffee and then complete questionnaires that relate to the PMT constructs. Intention and behaviour to drink alcohol will be compared between the two conditions over a 4-week period.

DETAILED DESCRIPTION:
According to Statistics Canada, over three-quarters of Canadians drink alcohol, with those aged 20 to 24 being the most likely to report drinking alcohol. The National Cancer Institute reports that there is strong evidence that alcohol drinking can cause several types of cancers and the consumption of alcoholic beverages is recognized as a known human carcinogen. The evidence shows that increased alcohol consumption, especially regular drinking over time, elevates the risk of developing alcohol-related cancers. Clear patterns have emerged between alcohol consumption and the development of colorectal cancer, with cases increasing particularly in young adults. With rising cases of alcohol-related cancers, particularly colorectal cancer in younger adults, and the widespread prevalence of alcohol consumption among this age group, this demographic becomes an important focus for preventative health strategies including targeted research and interventions. Therefore, the objective of the present study is to assess the effectiveness of an intervention grounded in the Protection Motivation Theory (PMT) to reduce alcohol-related intentions and behaviours among young Canadian adults. This study will provide valuable insights into young adults' drinking patterns and cancer awareness while supporting the development of effective interventions for reducing alcohol-related cancer risks in this vulnerable population. If the proposed intervention is successful, it can guide young adults into creating healthier habits and reduce the incidence and prevalence of colorectal cancer. Protection Motivation Theory (PMT) was introduced to explain the impact of persuasive communication on behaviour, with an emphasis on cognitive mechanisms underpinning the rationale to follow or not to follow a recommended behaviour. The framework outlines how threat and coping appraisals predict behavioural intentions, which then predict behaviour. Understanding the role that perceived vulnerability, perceived severity, response efficacy and self-efficacy of the PMT model play in affecting health behaviour change will help public health educators understand how to develop specific interventions to inform this population about the relationship between colorectal cancer and alcohol and enact positive change in the decision-making related to alcohol drinking.

This study will be a two-armed randomized control trial (RCT) with repeated measures (i.e., baseline, post-intervention, and 4-week follow-up). Participants will be randomly allocated to treatment groups using block randomization and a random number generator to place participants in groups of two (intervention and attention control). The block randomization method will be conducted following the Student Investigator (SI) acquiring consent and the LOI form. Participants will then be provided with their specific study number via email. Participants will be recruited through a variety of avenues: through the Mass Recruitment system at Western University, through Facebook groups, and presentations at university club meetings and classes. Posters will be displayed across the Western campus and London and lastly through informal conversation between peers. All recruitment aids will inform the interested participant to contact the SI to receive the information letter. The PMT intervention group will be given a video podcast relating to the threat and coping appraisal components of PMT (perceived severity, perceived vulnerability, response-efficacy and self-efficacy) and include information pertaining to alcohol and its correlation to colorectal cancer. The attention control group will also be given a video podcast, however, this video will focus on general information about coffee instead of specific alcohol and colorectal cancer information. This study will be conducted entirely online, with no in-person components for participants. Upon enrollment, participants will be provided with a Letter of Information (LOI) to review, electronically sign, and submit via email. At baseline, participants will be required to complete a series of surveys that assess their drinking patterns, drinking intentions, Protection Motivation Theory (PMT) constructs, and demographic information via Qualtrics. After submitting this baseline data, one week later, participants will receive a podcast video link via YouTube. The PMT intervention video podcast will be created using iMovie on MacOS and will be a 7-minute informational video explaining the current research on alcohol and its relationship to colorectal cancer and colorectal cancer risks associated with alcohol. This will be within the context of both the threat and coping appraisals of the PMT that highlights the severity of colorectal cancer, the susceptibility of colorectal cancer and the efficacy of a coping response to reduce alcohol consumption., while those in the attentional-control group will receive general information about coffee. Following the video, participants will be asked to immediately complete surveys on the PMT constructs and their alcohol-related intentions. At the final time point, 4 weeks post-intervention, participants will be asked to complete the same surveys again, including those assessing PMT, intentions, and actual drinking behaviour. All study materials, including links to the surveys, will be sent to participants via the email address they provided at the start of the study to the SI.

The primary objectives of this study are to investigate whether the use of an informational video linking alcohol use and colorectal cancer, following the threat and coping appraisal components of the Protection Motivation Theory (PMT) framework, reduces alcohol drinking intention and behaviour among young Canadian adults. Additionally, we are aiming to determine whether perceived vulnerability, perceived severity, response efficacy and self-efficacy are associated with goal intentions to reduce drinking alcohol and whether goals intentions to reduce drinking alcohol are associated with actual reductions in alcohol use. Threat and coping appraisals, goal intention and behaviour will be assessed using online self-report questionnaires at baseline, immediately post-intervention and 4 weeks through Qualtrics. We hypothesize that those exposed to the threat and coping appraisal information grounded in the PMT components of severity, vulnerability, response efficacy, and self-efficacy will achieve higher scores on purpose-built questions reflecting these components compared to their control counterparts focused on attentional information. We further hypothesize that those exposed to the threat and coping appraisal information grounded in the PMT components of severity, vulnerability, response efficacy and self-efficacy will show lower intentions to drink alcohol and lower alcohol use compared to their attentional information control counterparts. Finally, we hypothesize that increases in severity, vulnerability, response efficacy and self-efficacy of alcohol usage will be associated with a reduction in intentions to drink. Data collected throughout this study will be quantitative in nature and will be analyzed using a variety of statistical tests which could include t-tests, analysis of variance, correlation analyses, and multiple regression analyses. Descriptive statistics will be done and continuous data will be presented with standard deviation, mean, median and range. As data will be collected at multiple points throughout the study, a repeated measures analysis will be used to analyze the outcomes of variables at different points throughout the study. This will allow for the comparison between the intervention and control groups as the repeated measures correlation model tells us the strength of the linear correlation between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19-25 Able to read, write and understand English
* Current alcohol drinker
* Access to necessary resources for a technology-based intervention (i.e., smartphone, computer, internet)

Exclusion Criteria:

* Under the legal drinking age in Ontario of 19 at the time of signing the consent form
* Currently actively participating in behaviour therapy treatment for alcohol or attending a rehab centre
* Are pregnant /plan to become pregnant during the study period

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol Intention | From enrollment to the end of treatment at 4-weeks post-intervention.
  Participants alcohol intentions measured using an online questionnaire.
Alcohol Behaviour | From enrollment to the end of treatment at 4-weeks post-intervention.
  Participants alcohol consumption as measured using an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Parapavessis, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Drinking Among Young Adults — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6876515/
- See also: Efficacy of a non-drinking mental simulation intervention for reducing student alcohol consumption — https://journals-scholarsportal-info.proxy1.lib.uwo.ca/pdf/1359107x/v20i0004/688_eoanmsifrsac.xml_en
- See also: Colorectal Cancer in Young People — https://www.yalemedicine.org/news/colorectal-cancer-in-young-people
- See also: Protection Motivation Theory (PMT) — https://open.ncl.ac.uk/theories/10/protection-motivation-theory/
- See also: Alcohol and Cancer Risk — https://www.cancer.gov/about-cancer/causes-prevention/risk/alcohol/alcohol-fact-sheet